## Effect of tDCS on Cognition, Symptoms in Chronic Schizophrenia Patients With Tardive Dyskinesia

V1.0 2017.06.01

NCT03497013 Research Report Table

| Name of the Research Center: | |
|------------------------------|--------------|
| Name of the Research doctor: | |
| Name abbreviation: | <u> _ _ </u> |
| No.: | |

## **Guidance Notes for the Subjects**

**(Brief introduction)** This research is a mandatory project of Suzhou Science and Technology Bureau, which is undertaken by Suzhou Psychiatric Hospital (Project No. SS201752). At present, it has imported tDCS, a new method of brain stimulation therapy, which is a new method in the world, and associated with CANTAB and other evaluation tools of objective monitoring. At the same time, it was used for the genetic testing to explore the efficacy and related mechanisms of schizophrenia with tardive dyskinesia.

【Check item】 1.tDCS treatment: it provides 15 treatment for you free of charge. 2. Clinical evaluation: a medical history collection, a clinical scale and a related questionnaire were conducted by the doctor to assess your clinical symptoms comprehensively, the seriousness of the disease, the improvement of symptoms, etc. 3. Genetic testing: it's needed to collect 5 ml of your venous blood for genetic examination.

**[Benefit and Risk]** If you meet the inclusion and exclusion criteria of the study, you will be subject to the above inspection. During the research period, you will be provided with free cognitive evaluation, clinical scale evaluation and genomics research, etc, and the corresponding subsidies will be given. You can keep abreast of the information data and research progress related to this research. During the study period, if you have any questions, you can contact the related people in this research group of this subject.

**[Participation principle]** It's your freedom that whether to participate in this research or whether to withdraw from it during the course of the study. It will not affect your follow-up treatment by refusing to participate in or withdraw from the study. If you need other treatments, or you don't follow the research plan, or you have a research related injury, or for any other reason, research physicians can terminate your continued participation in this study.

**Confidentiality** If you decide to participate in this research, your participation in the trial and the personal data in the trial are confidential. When the results of this study are published, it will not disclose any of your personal information.

## **Informed Consent of the Subjects**

I have read this informed consent.

I have a chance to ask and all the questions have been answered.

I understand that participation in this research is voluntary.

I can choose not to participate in this research, I won't be discriminated against or retaliated due to withdrawing after notify the researcher at any time, and my any medical treatment and rights and interests will not be affected for this.

If I need another treatment, or I don't follow the research plan, or there's any research related injury, or for any other reason, the research physician or researcher can terminate my continued participation in this study.

| study. | |
|---|---|
| Name of the subject: | Signature of the subject: |
| Date: | |
| I have accurately informed this docum | nent to the subjects, he / she has read the informed consent |
| accurately, and it proves that the subjects l | have the opportunity to ask questions. I certify that he / she is |
| voluntarily agreeing to it. | |
| Name of the researcher: | Signature of the researcher: |
| Date: | |